CLINICAL TRIAL: NCT01732445
Title: A Phase 2 Pilot Trial of Ruxolitinib Combined With Danazol for Patients With Primary Myelofibrosis (MF), Post Essential Thrombocythemia-Myelofibrosis (Post ET) and Post Polycythemia Vera Myelofibrosis (PV MF) Suffering From Anemia
Brief Title: Ruxolitinib Phosphate and Danazol in Treating Anemia in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC1283; NCI-2012-02201 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1283 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-05

CONDITIONS: Anemia; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Anemia; Primary Myelofibrosis | interventions — ruxolitinib; Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (ruxolitinib phosphate and danazol) (Experimental): Patients receive ruxolitinib phosphate PO BID and danazol PO TID on days 1-56. Treatment repeats every 56 days for 6 courses in the absence of disease progression or unacceptable toxicity. At the treating physician's discretion, patients may continue treatment past 6 courses if they are without disease progression.
  Interventions: Drug: ruxolitinib phosphate; Drug: danazol; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Drug: ruxolitinib phosphate — Given PO
  Other Names: INCB18424; Jakafi; oral JAK inhibitor INCB18424; oral Janus-associated kinase inhibitor INCB18424
Drug: danazol — Given PO
  Other Names: Chronogyn; DAN; Danocrine
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This phase II pilot trial studies how well ruxolitinib phosphate and danazol work in treating anemia in patients with myelofibrosis. Ruxolitinib phosphate and danazol may cause the body to make more red blood cells. They are used to treat anemia in patients with myelofibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy (best overall response) of ruxolitinib (ruxolitinib phosphate) and danazol in patients with myelofibrosis suffering from anemia.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival of patients with myelofibrosis suffering from anemia initiating ruxolitinib and danazol.

II. To evaluate the adverse event profile of ruxolitinib and danazol in patients with myelofibrosis suffering from anemia.

TERTIARY OBJECTIVES:

I. To evaluate quality of life (QOL) and patient-reported symptoms using the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) and European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) with ruxolitinib and danazol for patients with myelofibrosis suffering from anemia.

OUTLINE:

Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) and danazol PO thrice daily (TID) on days 1-56. Treatment repeats every 56 days for 6 courses in the absence of disease progression or unacceptable toxicity. At the treating physician's discretion, patients may continue treatment past 6 courses if they are without disease progression.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of primary myelofibrosis (MF), post polycythemia vera (PV) or post essential thrombocythemia (ET) myelofibrosis (intermediate 1, intermediate II or high risk) requiring medical therapy
* Anemia is required for trial entry (defined as hemoglobin < 10g/dL or transfusion dependent [having needed a transfusion anytime in the past 6 months])
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at study entry
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 50,000/uL
* Serum creatinine =< 1.5 x the upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN; if total bilirubin is > 1.5 x ULN, a direct bilirubin should be performed and must be < 1.5mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN; higher values (i.e., =< 5 x ULN) are allowed if clinically compatible with hepatic extramedullary hematopoiesis
* Life expectancy of >= 6 months
* Patient able to provide voluntary written informed consent to participate
* Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria:

* Any chemotherapy (e.g., hydroxyurea), immunomodulatory drug therapy (e.g., thalidomide, interferon-alpha), immunosuppressive therapy, corticosteroids > 10 mg/day prednisone or equivalent, or growth factor treatment (e.g., erythropoietin), hormones (e.g., androgens, danazol) =< 14 days prior to registration; note: patients who are on ruxolitinib may continue on without a 14 day wash out at the treating physician's discretion
* Major surgery =< 28 days or radiation =< 6 months prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Active acute infection requiring antibiotics
* Uncontrolled congestive heart failure (New York Heart Association classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass, graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to registration
* Participation in any study of an investigational agent (drug, biologic, device) =< 30 days, unless during non-treatment phase
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness
* Clinically active hepatitis B or C
* Active malignancy other than MF, except adequately treated basal cell carcinoma and squamous cell carcinoma of the skin, cervical carcinoma in situ or other malignancies that have been stable and off therapy for 5 years
* Patient currently taking simvastatin, or lovastatin at a dose greater than 10 mg/day
* Men with prostate specific antigen (PSA) > 4 ng/ml or with uncontrolled benign prostatic hypertrophy
* Patient received prior combination treatment with ruxolitinib and danazol together; note: previous treatment with ruxolitinib and/or danazol as single agent therapy is allowed
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); use of the following strong or moderate inhibitors are prohibited =< 7 days prior to registration

  * Strong inhibitors of CYP3A4:

    * Indinavir (Crixivan)
    * Nelfinavir (Viracept)
    * Atazanavir (Reyataz)
    * Clarithromycin (Biaxin, Biaxin XL)
    * Itraconazole (Sporanox)
    * Ketoconazole (Nizoral)
    * Nefazodone (Serzone)
    * Saquinavir (Fortovase, Invirase)
    * Telithromycin (Ketek)
  * Moderate inhibitors of CYP3A4

    * Erythromycin (Erythrocin, E.E.S., Ery-Tab, Eryc, EryPed, PCE)
    * Fluconazole (Diflucan)
    * Grapefruit juice
    * Verapamil (Calan, Calan SR, Covera-HS, Isoptin SR, Verelan)
    * Verelan PM
    * Diltiazem (Cardizem, Cardizem CD, Cardizem LA, Cardizem SR, Cartia XT, Dilacor XR, Diltia XT, Taztia XT, Tiazac)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Mesa, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Tisch Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care (Ruxolitinib Phosphate and Danazol): Patients receive ruxolitinib phosphate PO 10 mg BID and danazol PO 200 mg TID on days 1-56. Treatment repeats every 56 days for 6 courses in the absence of disease progression or unacceptable toxicity. At the treating physician's discretion, patients may continue treatment past 6 courses if they are without disease progression.
Period: Overall Study
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 70.5 [43 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate as Determined by International Working Group Criteria
Description: Best overall response rate as determined by International Working Group criteria: An evaluable patient will be classified as a responder for the primary endpoint if the patient's best overall response is CR, PR or CI (Clinical Improvement) as determined by International Working Group Criteria over all cycles of study treatment. The percentage of successes will be estimated by the number of successes (defined as complete response, partial response, or clinical improvement) divided by the total number of evaluable patients times 100. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients with CR, PR or CI
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Number analyzed (Participants) | 14
percentage of patients with CR, PR or CI | 28.6 [8.4 to 58.1]

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier. The median and 95% confidence interval are reported below.
Time Frame: From registration to death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Number analyzed (Participants) | 14
months | 19.2 [4.1 to 28.8]

3. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Number analyzed (Participants) | 14
percentage of patients
  Platelet count decreased | 7.1
  Anemia | 64.3
  White blood cell decreased | 7.1
  Neutrophil count decreased | 14.3
  Hypertension | 7.1
  Premature menopause | 7.1

4. Other Pre Specified Outcome: Patient-reported Symptoms Assessed Using the MPN-SAF, as Measured by the Percentage of Patients With a Decrease in MPN-SAF TSS Greater Than 50% From Baseline
Description: Patient-reported symptoms will be described at each time point using the mean, confidence interval, median, and range. The Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) will be analyzed using published scoring algorithms. MPN-SAF includes 27 items scored on a scale of 0 to 10. The MPN-SAF Total Symptom Score (TSS) (range 0-100) was computed according to the published scoring algorithm. Higher scores represent worse symptom burden. The percentage of patients with a decrease in MPN-SAF TSS greater than 50% from baseline and 95% confidence interval are reported below.
Time Frame: Baseline to up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
Number analyzed (Participants) | 14
percentage of patients | 28.6 [8.4 to 58.1]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Supportive Care (Ruxolitinib Phosphate and Danazol)
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Ruxolitinib Phosphate and Danazol) (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Ruxolitinib Phosphate and Danazol) (N=14)
Anemia (Blood and lymphatic system disorders) | 9 (24)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 3 (6)
Edema limbs (General disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 12 (29)
White blood cell decreased (Investigations) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes